CLINICAL TRIAL: NCT05991063
Title: The Ability Of Inferior Vena Caval Distensibility Index With Passive Leg Raising Test To Predict Spinal Anesthesia-induced Hypotension In Elderly Patients Undergoing Infra-umbilical Surgeries. A Prospective Observational Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdelghany ali, Lecturer of anesthesia, Cairo University
Other Study IDs: Ms2022
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Spinal Anesthetics Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many previous studies have investigated the ability of various methods such as passive leg raising test , and inferior vena cava collapsibility index in predicting post-spinal hypotension, but none of them have succeeded in obtaining a good predictive value.

Our study aims to combine the passive leg raising test with the inferior vena cava distensibility index to aid in predicting post-spinal hypotension in elderly undergoing infra-umbilical surgeries.

ELIGIBILITY:
Inclusion Criteria:

* 1. 65 years of age or more. 2. ASA score I & II. 3. Patients are scheduled for infra umbilical surgeries under spinal anesthesia.

Exclusion Criteria:

* Negative consent. Pre-existing hypertension Diabetes mellitus or autonomic neuropathy (patients diagnosed with autonomic neuropathy or having suggestive symptoms such as orthostatic hypotension, syncopal attacks, decreased sweating, and urinary incontinence) Emergency operations Absolute contraindications or failure to perform spinal anesthesia If PLR maneuver is contraindicated (intracranial hypertension) or possibly unreliable ( venous compression stocking, intraabdominal hypertension) Difficulties in IVC visualization due to increased subcutaneous fat tissue or gastric gas interferin

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A total of 68 consecutive elderly patients, aged >65 years scheduled for elective infra-umbilical surgical operations under spinal anesthesia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of Δmax.IVCd in predicting post-spinal anesthesia hypotension in elderly patients. | 15 minutes before spinal anesthesia
  The incremental changes of measured maximum inferior vena caval diameter after passive leg raising